CLINICAL TRIAL: NCT05988151
Title: New Surgical Approach in Labioplasty: Inspired by the Fibonacci Ratio
Brief Title: New Surgical Approach in Labioplasty
Status: Completed | Type: Observational
Sponsor: Batman Training and Research Hospital (Other Government)
Responsible Party: Principal Investigator, Erhan Okuyan,M.D, M.D Obstetrics and Gynecology specialist, Batman Training and Research Hospital
Other Study IDs: 2022/25
Record Dates: First submitted 2023-08-04; First posted 2023-08-14 (Actual); Last update posted 2023-10-17 (Actual); Status verified 2023-10

CONDITIONS: Gynecologic Disease; Surgery-Complications
Keywords: Labioplasty; Vaginoplasty; Fibonacci ratio
MeSH Terms: conditions — Genital Diseases, Female

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- New surgical approach (Fibonacci ratio): Agroup of 60 patients who underwent VaGinoplasti+ labioplasty ( wedge resection) with fibonacci ratio surgical ratio.
  Interventions: Other: New surgical approach
- Classical surgical approach (control group): A group of 30 patients who underwent Vaginoplasty + Labioplasty( wedge resection) with classical surgical approach.

INTERVENTIONS:
Other: New surgical approach — Patients were included in the study after obtaining informed consent for the new surgical approach inspired by the Fibonacci ratio.
  Groups: New surgical approach (Fibonacci ratio)

SUMMARY:
The data of patients who underwent labiaplasty + vaginoplasty between 2020 and 2022 by a single surgeon in our clinic were analyzed. Preoperative and postoperative FSFI (Female sexual function index) questionnaire scores were used to compare the results of the classical surgical approach and the new surgical approach technique designed according to the Fibonacci ratio in the early postoperative period such as operating time, bleeding amount, etc.

DETAILED DESCRIPTION:
The data of patients who underwent labiaplasty + vaginoplasty between 2020-2022 for reasons such as vaginal laxity, personal hygiene problems, recurrent vaginal infections were analyzed retrospectively. The data of the patients who underwent fibonacci ratio, which is a new surgical approach technique( by Okuyan E. M.D), and the patients who underwent classical surgical technique were taken from their files and retrospectively analyzed. Data including age, body mass index, number of live births, preoperative FSFI, FGSIS and postoperative one month FSFI (Female sexual function index) and FGSIS (The Female Genital Self-Image Scale) scores were recorded and compared between both groups.

ELIGIBILITY:
Inclusion Criteria:

1. No history of any disease
2. The presence of at least 2 of the reasons such as dislike of cosmetic appearance, vaginal abundance, personal hygiene disorder, difficulty in wearing underwear.
3. Body mass index between 15-25
4. Informed consent has been obtained for the new surgical approach technique.
5. Not taking any medication continuously
6. Willing to participate in the study.

Exclusion Criteria:

1. Absence of at least 2 of the reasons such as dislike of cosmetic appearance, vaginal

   abundance, personal hygiene disorder, difficulty in wearing underwear.
2. History of continuous medication, alcohol and/or smoking.
3. History of chronic diseases (Asthma, Diabetes mellitus, Cardiac disease, Psychiatric disease etc.)
4. Body mass index outside the range of 15-25.
5. Not wanting to be included in the study or wanting to leave the study after inclusion.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Study Population: Patients who underwent labioplasty plus vajinoplasti prosedures in our clinic (age 18-45 years old)
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2022-04-12 (Actual); Primary Completion 2023-07-01 (Actual); Study Completion 2023-08-02 (Actual)

PRIMARY OUTCOMES:
To be able to standardize genital harmony using fibonacci ratio. | Postoperative 1 month
  To standardize the genital harmony with a holistic approach with the Fibonacci ratio with a purely mathematical ratio outside the existing classification systems (in contrast to Banwell, Motakeff classifications).

SECONDARY OUTCOMES:
To adapt the fibonacci ratio to female genital cosmetic surgery | Postoperative 1 month
  To adapt the fibonacci ratio applied in breast and facial aesthetics to female genital aesthetic surgery procedures.

CONTACTS AND LOCATIONS:
Overall Officials: Erhan Okuyan, Principal Investigator — Batman Training and Research Hospital
Locations (1):
- Batman Training and Research Hospital, Batman, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Share after publication